CLINICAL TRIAL: NCT03244969
Title: Study of the Granulation Tissue Formation in the Early Fracture Hematoma
Brief Title: Bone Healing Study
Status: Withdrawn | Type: Observational
Why Stopped: Study was registered in another clinicaltrials.gov entry
Sponsor: Kazan Federal University (Other)
Responsible Party: Principal Investigator, Mikhail Mavlikeev, aspirant of the morphology department, Kazan Federal University
Other Study IDs: hematoma-2017
Record Dates: First submitted 2017-08-07; First posted 2017-08-10 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Bone Fracture
Keywords: Hematoma fracture, angiogenesis, bone formation
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the research is to identify structural tissue changes in the early fracture hematomas.

DETAILED DESCRIPTION:
The fracture hematomas obtained during reconstructive bone surgery from patients with bone fractures will be examined. Histological methods and ultra-thin sections for electron microscopy will be used to identify structural tissue changes in the granulation tissue in different period of time after bone fracture. Immunohistochemical analysis will be performed to estimate the dynamic of proliferation, differentiation and cell migration during granulation and reticulofibrosis bone tissues development.

ELIGIBILITY:
Inclusion Criteria:

* Patients with fractures of the upper and lower extremities
* Patients for whom the surgical bone reconstruction are indicated

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with fractures of the upper and lower extremities underwent surgical bone recunstruction.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-10 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Granulation tissue formation | 23 days

CONTACTS AND LOCATIONS:
Locations (1):
- Igor Plaksa, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes